CLINICAL TRIAL: NCT04376424
Title: Hand Carried Ultra-Sound Assisted Medical Management of Acute Decompensated Heart Failure. A Randomized Controlled Trial (USA-HF)
Brief Title: Ultra-sound Assisted Management of Heart Failure
Acronym: USA-HF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No data has been collected, no subjects enrolled
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-0276
Record Dates: First submitted 2020-04-14; First posted 2020-05-06 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Ultra Sound Guided Therapy Group (Experimental): Hand carried ultrasound will be used in this group to measure IVCd, collapsibility along with internal jugular vein collapsibility. The results of the ultrasound will be unblinded to the treating team.
  Interventions: Diagnostic Test: Hand Held Ultrasound
- Conventional Therapy Group (No Intervention): Conventional therapy will occur the use of hand carried ultrasound. The results will be blinded to the treating team. The managing team will analyze the data at the end of the study.

INTERVENTIONS:
Diagnostic Test: Hand Held Ultrasound — Guideline directed medical therapy for heart failure with the addition of hand held ultrasound
  Arms: Ultra Sound Guided Therapy Group

SUMMARY:
The purpose of this study is to evaluate the impact of using hand carried ultrasound measurements of volume status in directing treatment of heart failure patients admitted with acute exacerbation.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of using hand carried ultrasound measurements of volume status in directing treatment of heart failure patients admitted with acute exacerbation. The use of hand carried ultrasound is expected to reduce hospital Length of stay, heart failure re-admission rates, emergency room visits and in hospital complications such as renal failure. The hypothesis tested is as follows:

Null: The use of hand carried ultrasound in the management of heart failure patients did not change outcome.

Alternative: The use of hand carried ultrasound in the management of heart failure patients did change outcome.

The study endpoints are as follows:

1. A primary endpoint will be the impact of using hand carried ultrasound on length of hospital stay.
2. The secondary endpoint will be 30 days re-admission following heart failure hospitalization, emergency room visits and in hospital complications such as renal failure.

This is a randomized controlled un-blinded study that poses very minimal risk because patients will only undergo an ultrasound measurement of Inferior vein cava (IVC) and internal jugular vein diameter and compressibility. Also, the society will benefit greatly with the prospect of reducing hospitalization and medical complications, optimizing healthcare delivery to heart failure patients, and reducing hospitalization cost. The results of this study/study procedure will only direct medical therapy that heart failure patients usually receive through routine care such as dose and frequency of diuresis.

ELIGIBILITY:
Inclusion Criteria:

1. New admission from emergency department to heart failure ( red team) service for acute exacerbation of heart failure ( defined based on clinical and imaging characteristics , shortness of breath due to volume overload, CXR showing pulmonary vascular congestion/pulmonary edema, elevated NTproBNP, dyspnea Not secondary to infectious process (pneumonia).
2. Heart failure NYHA class III, IV
3. Age>=18 years old

Exclusion Criteria:

1. End stage Renal disease on dialyses (ESRD on HD) or stage V CKD (defined as GFR<15)
2. end stage Heart failure on chronic inotrope (example Milrinone)
3. Renal failure that deemed to be secondary to other reason (dehydration, renal or post renal (obstructive)
4. morbid obesity BMI > 40
5. incarcerated patients (prison) TDC.
6. pregnant patients
7. Patients with dyspnea not mainly due to heart failure, ESRD patients, intubated patients
8. Aged less than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
length of hospital stay (days) | Immediately after discharge
  number of days from admission to discharge

SECONDARY OUTCOMES:
Number of participants readmitted for heart failure with 30 days of discharge, and percentage of participant out of all participants in each group readmitted in each group within 30 days | One month after discharge
  Follow up telephone call after discharge
number of participant readmitted for any reason within 30 days of discharge, and percentage of participant ( out of all participant in each group) readmitted in each group within 30 days of discharge. | One month after original discharge
  assessment of readmission to hospital
percent change in GFR | One month after original discharge
  amount of change in GFR
hospitalization Cost | immediately after discharge of hospitalization
  hospitalization cost measured for all hospitalization stay from admission to discharge for each participant
Time to readmission | assessed within 4 weeks from index admission (i.e. thirty days readmission)
  time between original hospitalization and readmission
Number of right heart catheterization in each group and percentage of right heart catheterization in each group | One month after admission
  document what procedures were done

CONTACTS AND LOCATIONS:
Overall Officials: Wissam Khalife, MD, Principal Investigator — University of Texas Medical Branch Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No